CLINICAL TRIAL: NCT02368132
Title: Comparative Effectiveness of Delivery Methods for Caregiver Support and Education
Brief Title: Delivery Models of Caregiver Support and Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 14-080; 01548 (Other: IRB)
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Dementia
Keywords: Caregivers; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): Caregivers randomized to UC will be sent general material about VA and community resources for patients with dementia and their CGs. With the exception of this material, individuals in this group will receive usual care and will be contacted again at 3, 6, and 12 months for follow-up research assessments.
- Individual Delivered TEP Arm (Active Comparator): Two mandatory modules that cover the stages of dementia and provide a brief introduction to problem solving techniques, action plan development, and coping skills, plus a menu of additional modules covering various content areas evaluated during the course of the monthly assessments (e.g., communication skills, behavioral management techniques, stress management and coping skills, longterm planning, etc.). Each individual TEP session will begin with reviewing education related to the selected module. The remainder of each session will involve coaching the caregiver on emotion-focused and problem focused coping strategies. The care manager will also discuss problem solving with the CG to reinforce the action plan and the educational component of the intervention.
  Interventions: Behavioral: Individual Delivered TEP
- Group Delivered TEP Arm (Active Comparator): All TEP modules will be in a group format. Each call will take 1.5-2 hours. Each group will be comprised of 5-8 CGs who will call into a teleconference line at a pre-specified time. Groups will include spouse/partner-only or adult child-only CGs. The content of the calls will mirror those in the individual TEP delivered program. In addition to the group calls, they will receive individual care management.
  Interventions: Behavioral: Group Delivered TEP

INTERVENTIONS:
Behavioral: Group Delivered TEP — All TEP modules will be in a group format. Each call will take 1.5-2 hours. Each group will be comprised of 5-8 CGs who will call into a teleconference line at a pre-specified time. Groups will include spouse/partner-only or adult child-only CGs. The content of the calls will mirror those in the individual TEP delivered program. In addition to the group calls, they will receive individual care management.
  Arms: Group Delivered TEP Arm
Behavioral: Individual Delivered TEP — Two mandatory modules that cover the stages of dementia and provide a brief introduction to problem solving techniques, action plan development, and coping skills, plus a menu of additional modules covering various content areas evaluated during the course of the monthly assessments (e.g., communication skills, behavioral management techniques, stress management and coping skills, longterm planning, etc.). Each individual TEP session will begin with reviewing education related to the selected module. The remainder of each session will involve coaching the caregiver on emotion-focused and problem focused coping strategies. The care manager will also discuss problem solving with the CG to reinforce the action plan and the educational component of the intervention.
  Arms: Individual Delivered TEP Arm

SUMMARY:
The proposed study seeks to compare usual care and two different interventions for caregivers (CGs) of Veterans with dementia that are brief and administered by telephone. In the first intervention, care management (i.e., assistance from a nurse or social worker who works with the CG and Veteran's primary care providers), support, psychoeducation, and skills training are tailored to each individual CG and delivered on an individual basis. In the second intervention, care management is tailored and delivered to each individual CG, but support, psychoeducation, and skills training are delivered (also by phone) in a group format. This study will allow us to examine the added benefit of participating in a CG group that provides mutual peer support and feedback. The investigators also will evaluate the extent to which spousal vs. adult child CGs respond differently to the two interventions. Findings will help refine patient/CG-centered care management and support programs designed to facilitate access to services and improve the quality of life of Veterans with dementia and their families.

DETAILED DESCRIPTION:
Background: Existing interventions for informal caregivers (CGs) of care recipients (CRs) with dementia vary on multiple dimensions (e.g., content, administration time, mode of delivery), and findings indicate that these programs are effective in improving CG and CR outcomes. The investigators' team has developed and evaluated two CG programs that are unique in that they are relatively brief (i.e., 3 months) and rely solely on telephone administration. The original program, the Telehealth Education Program (TEP), provides CG support, psychoeducation, and skills training in a group format. The second program adapted the original TEP to be delivered to individual CGs and includes collaborative care management services. Key components of this CR/CG-centered program include direct collaboration among teams of care managers, primary care providers (PCPs), and CGs. The decision to develop an individually-tailored, collaborative care program was partly in response to the success of collaborative care models with other patient populations and the fact that the majority of individuals with dementia receive their healthcare from their PCPs. Nonetheless, an individually-delivered program lacks the benefits derived from the mutual peer support and feedback provided by group-based interventions. What remains to be determined, therefore, is whether modifying the individually-delivered care management program to deliver TEP in a group format is more effective than the individually-delivered program alone.

Objectives: The objectives of the project include: a) testing the comparative effectiveness of 2 delivery models (individual TEP + individual care management vs. group TEP + individual care management) of a telephone-based, collaborative dementia care intervention for CGs, and b) exploring whether the individual or individual + group intervention is more effective/acceptable among spousal vs. adult children CGs.

Methods: To meet these objectives, the investigators will use a prospective, randomized control group, repeated measures (i.e., baseline, 3, 6, and 12 month follow-up) design. Participants will include 405 CGs (spouses and children 18 years of age and older) of Veterans diagnosed with dementia and receiving routine clinical care at two VA sites. CGs will be recruited for participation if they live with and/or provide 4+ hours of care/day. CGs will be randomly assigned to usual care, the individual intervention, or the individual + group intervention. The main objectives of both interventions are to facilitate resource connection and provide education, psychosocial support, and care management for individuals caring for Veterans with dementia, thereby improving access to and use of non-institutional services, rates of guideline adherent care, and CG/CR outcomes. In both interventions, CGs will receive education, continuous support, skills training, and monitoring of Veterans' medication adherence, symptoms, and service needs. CGs will be asked to complete an assessment battery of standardized measures of CR- and CG-characteristics. Veterans' clinical medical records (including cost data) also will be evaluated for screening and clinical data collection purposes. Generalized estimating equations (GEE) will be the primary method used to analyze the nested, longitudinal data.

ELIGIBILITY:
Inclusion Criteria:

* Veteran and CG are 18 years of age or older.
* Veteran is community dwelling.
* Veteran has had at least one PACT encounter at the Corporal Michael J. Crescenz VA Medical Center (CMCVAMC), VA Western New York Healthcare System (VAWNYHS), or affiliated community-based outpatient clinics in the past six months at the time that data is extracted from VINCI for recruitment.
* Veteran meets criteria for dementia that is verified by informant report (AD8, score of 2 or above).
* CG endorses that Veteran has a diagnosis of dementia.
* CG lives with or provides care for the Veteran for an average of at least 4 hours per day.
* Veteran's CG is willing and able to provide informed consent.
* CG is either a spouse/partner or adult child.
* CG screens positive for moderate CG burden (per Zarit Burden Interview (4-item) score of 3 or more).

Exclusion Criteria:

* CG cognitive, hearing, visual, or other physical impairments leading to difficulty with informed consent process, assessment, or participation in intervention visits.
* CG participation in a pre-existing support group or CG intervention at enrollment (however CGs can subsequently enroll in any treatment they choose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahrzad Mavandadi, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mavandadi S, Ingram E, Chen S, Klaus J, Oslin D. The association between social ties and changes in depressive symptoms among veterans enrolled in a collaborative depression care management program. Psychol Serv. 2022 Feb;19(1):111-117. doi: 10.1037/ser0000496. Epub 2020 Oct 8. PMID 33030946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregivers (CGs) of Veterans with dementia receiving primary care at the Corporal Michael J. Crescenz VA Medical Center, VA Western New York Healthcare System, and their affiliated outpatient clinics were recruited and enrolled between May 2016 and November 2019. Participants were sent a letter introducing them to the study following either direct provider referral or upon a review of lists of patients prescribed memory-enhancing medications generated from the electronic medical record.
Period: Overall Study
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm
Started | 112 | 122 | 85
Completed (3 Month Follow-Up Completed) | 32 | 71 | 50
Not Completed | 80 | 51 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm | Total
Number analyzed (Participants) | 112 | 122 | 85 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.31 (11.36) | 72.20 (11.45) | 71.42 (11.12) | 71.68 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 114 | 80 | 298
  Male | 8 | 8 | 5 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 23 | 15 | 62
  White | 81 | 89 | 69 | 239
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 6 | 8 | 1 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 122 | 85 | 319
Revised Memory and Behavior Problem Checklist (CG Reaction Score) [Mean (Standard Deviation); unit: score on a measure] — The Revised Memory and Behavior Problems Checklist (Reaction Subscale) measures CG distress in response to dementia-related symptoms. The RMBPC CG reaction subscale captured how bothered or upset CGs were in response to each endorsed dementia-related symptom (range=0-96, higher scores denote greater distress in response to symptoms)
  score on a measure | 16.23 (11.29) | 20.48 (14.17) | 17.88 (12.38) | 18.29 (12.83)
VR 12 - Mental Component Score [Mean (Standard Deviation); unit: score on a measure] — Perceived overall mental wellbeing were assessed with the Mental Component Score (MCS) subscale of the Veterans RAND 12-Item Health Survey (VR12). Higher scores denote greater mental wellbeing (range: 0-100)
  score on a measure | 48.45 (9.02) | 43.07 (11.38) | 45.88 (11.08) | 44.24 (11.32)
Zarit Burden Interview [Mean (Standard Deviation); unit: score on a measure] — The 12-item Zarit Burden Interview was administered to assess CGs' perceived caregiving burden (range=0-48, higher scores denote greater burden)
  score on a measure | 15.98 (7.40) | 20.29 (9.04) | 19.63 (9.09) | 18.63 (8.72)

OUTCOME MEASURES:

1. Primary Outcome: Revised Memory and Behavior Problems Checklist (Reaction Subscale)
Description: The Revised Memory and Behavior Problems Checklist (Reaction Subscale) measures CG distress in response to dementia-related symptoms. The RMBPC CG reaction subscale captured how bothered or upset CGs were in response to each endorsed dementia-related symptom (range=0-96, higher scores denote greater distress in response to symptoms)
Time Frame: 3 Months
Population: Intent-to-treat analysis included all randomized participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm
Number analyzed (Participants) | 112 | 122 | 85
score on a scale | 19.46 (1.97) | 14.31 (1.41) | 10.73 (1.65)
Statistical Analysis 1: Comparison: Usual Care vs Individual Delivered TEP Arm vs Group Delivered TEP Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least squares mean difference = -8.73, Standard Error of Mean 2.57 — Estimated difference in least square means between Usual Care (reference) and Group Delivered TEP arm at 3 months
Statistical Analysis 2: Comparison: Usual Care vs Individual Delivered TEP Arm vs Group Delivered TEP Arm; Test type: Superiority; p = 0.04, Mixed Models Analysis; Least squares mean difference = -5.15, Standard Error of Mean 2.42 — Estimated difference in least square means between Usual Care (reference) and Individual Delivered TEP arm at 3 months

2. Primary Outcome: Zarit Burden Interview (12 Item)
Description: The 12-item Zarit Burden Interview was administered to assess CGs' perceived caregiving burden (range=0-48, higher scores denote greater burden)
Time Frame: 3 Months
Population: Intent-to-treat analysis included all randomized participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm
Number analyzed (Participants) | 112 | 122 | 85
score on a scale | 16.66 (1.25) | 17.95 (0.93) | 17.37 (1.09)

3. Primary Outcome: Veterans RAND 12-Item Health Survey (VR12)
Description: Perceived overall mental wellbeing were assessed with the Mental Component Score (MCS) subscale of the Veterans RAND 12-Item Health Survey (VR12). Higher scores denote greater mental wellbeing (range: 0-100)
Time Frame: 3 Months
Population: Intent-to-treat analysis included all randomized participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm
Number analyzed (Participants) | 112 | 122 | 85
score on a scale | 49.28 (1.52) | 45.29 (1.11) | 46.20 (1.32)

ADVERSE EVENTS:
Time Frame: Up to 1 year following baseline assessment
Arm/Group | Usual Care | Individual Delivered TEP Arm | Group Delivered TEP Arm
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/122 | 0/85
Serious Adverse Events (participants affected / at risk) | 3/112 | 7/122 | 6/85
Other Adverse Events (participants affected / at risk) | 0/112 | 0/122 | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=112) | Individual Delivered TEP Arm (N=122) | Group Delivered TEP Arm (N=85)
Hospitalization due to surgery (General disorders) | 1 (1) | 2 (2) | 3 (3)
Hospitalization - Illness (General disorders) | 2 (2) | 1 (1) | 1 (1)
Hospitalization/ER (General disorders) | 0 (0) | 3 (3) | 0 (0)
Surgery (General disorders) | 0 (0) | 1 (1) | 2 (2) — outpatient

LIMITATIONS AND CAVEATS:
Significant sample attrition precluded the ability to run comparisons beyond the three month follow-up or more complex interaction models.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02368132/Prot_SAP_000.pdf